CLINICAL TRIAL: NCT04645485
Title: A Phase 1 Study Evaluating the Safety and Tolerability of Autologous Non-hematopoietic Peripheral Blood Stem Cells Therapy in Healthy Adult Volunteers in Abu Dhabi, 2020 (SANTANA Study).
Brief Title: Safety and Tolerability of Autologous Non-hematopoietic Peripheral Blood Stem Cells Therapy in Healthy Adult Volunteers.
Acronym: SANTANA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abu Dhabi Stem Cells Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT.002.1.0.SANTANA
Record Dates: First submitted 2020-11-21; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: Nebulization; Autologous non-hematopoietic peripheral blood stem cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Nebulization of autologous non-hematopoietic peripheral blood stem cells (NHPBSC).
  Interventions: Biological: Nebulization of autologous non-hematopoietic peripheral blood stem cells (NHPBSC).

INTERVENTIONS:
Biological: Nebulization of autologous non-hematopoietic peripheral blood stem cells (NHPBSC). — Participants received the investigational therapy through compressor (jet) nebulization, in two doses divided on Days 0 and 1. Each dose contains 10 mL of peripheral blood-derived stem cells CD45-/CD90+/CD133+.
  Other Names: UAECell19

SUMMARY:
SANTANA Study is a phase 1, prospective, monocentric, open-label clinical trial involving healthy adult volunteers, with the objective to evaluate the safety and tolerability of the compressor nebulization of autologous non-hematopoietic peripheral blood stem cells (NHPBSC).

DETAILED DESCRIPTION:
The study was conducted in Abu Dhabi Stem Cells Center (ADSCC), and the cell processing and investigational product formulation were performed at the same center according to Good Laboratory Practices (GLPs) and Good Manufacturing Practices (GMPs). Participants received the investigational therapy through compressor (jet) nebulization (two doses divided on Days 0 and 1). The primary endpoint was the safety assessment, to be measured as Adverse Reactions (ARs) incidence [by the World Health Organization - Uppsala Monitoring Centre (WHO-UMC) causality assessment system], and the nebulization tolerability rate (Days 0 and 1). The Laboratory testing profile was evaluated before treatment (Day 0 or -1) and on Days 14 and 28. Two thorax radiography tests (chest X-rays - CXR) were assessed: before the therapy (Day 0 or -1) and on Day 7. An electrocardiogram (ECG) assessment was performed on Days 0 (or -1), 14, and 28. The application of the validated St. George's Respiratory Questionnaire (SGRQ) on Days 0 and 28 was a surrogate safety endpoint. The whole clinical assessment in SANTANA Study was daily recorded until Day 28, taking into account the ARs incidence. The secondary endpoint was the tolerability assessment, measured by nebulization tolerability rate (Days 0 and 1), and Adverse Events (AEs) tolerability within 28-days. The trial was approved by the ADSCC Research Ethics Committee, and written informed consent was obtained from all participants. SANTANA Study was conducted following the Declaration of Helsinki principles and Good Clinical Practices (GCPs), and the authors are responsible for designing the trial, compiling, and analyzing the data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female volunteers (18-50 years inclusive). Healthy subjects: volunteers not having any mental or physical diagnosed disorder or requiring regular or frequent medication, who is not known to suffer any significant illness, who should be within the ordinary range of body measurements)
* Non-smoking volunteers, based on self-reporting who have not used tobacco or nicotine-containing products (or less than 100 cigarettes or equivalent in his / her lifetime), including commercially available cigarettes, hand-rolled cigarettes, bidis, cigars, chewing tobacco, pipes, hookahs, shishas, snuff, snus, electronic cigarettes and similar devices, and nicotine replacement therapy within the last 12 months.
* Body mass index (BMI) ≥ 19 kg/m².
* For females: premenopausal, non-lactating, and non-pregnant.
* Ability to comply with test requirements and peripheral blood stem cell collection.
* The subject agrees to participate in the study and signs the SANTANA Study informed consent form.

Exclusion Criteria:

* Pediatric subjects (aged < 18 years) or older than 50 years' volunteers.
* Any clinically relevant gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, urological, immunological, and cardiovascular diseases or any other condition including clinically significant abnormal Laboratory parameters that, in the opinion of the Investigator, could jeopardize the safety of the subject.
* Current smoking subjects (or former smokers who have quit smoking three months before eligibility assessment).
* Body mass index (BMI) < 19 kg/m².
* For females: Postmenopausal, lactating or pregnant women.
* Donation or receipt of whole blood or blood products within three months before the screening visit.
* Inability to comply with test requirements or peripheral blood stem cell collection.
* Organ or cell transplants in the past three months.
* History of malignancies in the past five years.
* Have participated in other clinical trials in the past three months.
* Employee of Abu Dhabi Stem Cells Center (ADSCC) or their first-degree relatives (parent, sibling, or child).
* Inability to provide informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Adverse reactions (AR) incidence. | Days 0-28.
  Proportion of participants with treatment-related adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 and the WHO-UMC system for the causality assessment.
St. George's Respiratory Questionnaire (SGRQ) scoring. | Days 0, 28.
  Assessment of scoring changes.
Nebulization tolerability rate. | Days 0, 1.
  Proportion of participants that tolerate the NHPBSC nebulization successfully.
Adverse Events (AEs) tolerability rate. | Days 0-28.
  Proportion of participants that tolerate AEs -if any, and finish the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Abu Dhabi Stem Cells Center, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No